CLINICAL TRIAL: NCT05119582
Title: High-Intensity Focused Ultrasound (HIFU), a Novel Method for Treatment of Cutaneous Neurofibromas in Neurofibromatosis Type 1: Safety and Efficacy
Brief Title: HIFU Treatment of Cutaneous Neurofibromas in Neurofibromatosis Type 1: Safety and Efficacy
Acronym: cNF-HFU2101
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Joergen Serup (Other)
Collaborators: Sahlgrenska University Hospital (Other)
Responsible Party: Sponsor-Investigator, Joergen Serup, Professor, Chief Physician, Department of Dermatology, Bispebjerg Hospital
Organization: Bispebjerg Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIV-21-09-037759
Record Dates: First submitted 2021-10-29; First posted 2021-11-15 (Actual); Results first posted 2024-10-16 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-07

CONDITIONS: Cutaneous Neurofibroma

STUDY DESIGN:
Intervention Model Description: The study is a multicenter (two-center) open-label study with high-intensity focused ultrasound (HIFU) treatment of patients with the genetic disease Neurofibromatosis Type1.
  The study is not comparative or randomized. The investigation is performed prior to CE mark to confirm safety and performance of the System ONE-M device when used as intended, i.e. as an non-invasive method to remove cutaneous neurofibromas by 20 MHz high intensity focused ultrasound.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TOOsonix System ONE-M (Experimental): Cutaneous neurofibromas will be treated by high intensity focused ultrasound.
  Interventions: Device: TOOsonix System ONE-M

INTERVENTIONS:
Device: TOOsonix System ONE-M — Selected neurofibromas will be treated by high intensity focused ultrasound. Untreated fibromas will be used for controls.

SUMMARY:
The overall objective is to demonstrate safety and efficacy of HIFU treatment of cutaneous neurofibromas located close to the surface of the skin in patients with the genetic disease Neurofibromatosis Type 1. The study will use a new investigational equipment that has been specially developed for dermatological therapy.

The study includes 20 patients in total distributed between the two centers, each having a minimum of 8 cutaneous neurofibromas eligible for treatment. All participants are adults (over 18 years) of both sexes.

The new treatment method is based on focusing intensive ultrasound just below the skin surface. This creates a very fast localized heating in small and very well-defined volumes containing neurofibroma tissue. This heating destroys or weakens the tissue, and the body's natural processes will subsequently transport affected cells away through the lymphatic and vascular systems. During the healing-process, the rejected tissue is replaced by new skin cells that are not expected to be fibrous.

The treatment is intended to be carried out without breaking the skin surface, and open wounds are therefore avoided. This is an essential advantage of the method compared to all existing therapies, which are based on physical removal of tumors through an open skin surface (e.g. surgery or laser therapy). Complications with risk of pain, infection and scarring will therefore be significantly reduced with the new proposed method.

The treatment is carried out by sending focused ultrasound from the handpiece of the equipment into the target area with neurofibromas. The equipment is set to send doses of approximately 150 milliseconds (0.15 seconds). The skin area and HIFU doses can be followed on the system computer screen and will be placed side-by-side with approximately 1-2 millimeter spacing. To achieve good energy transfer from handpiece to skin, ordinary ultrasound gel is used. There are no other special pre-treatments or preparations for the process. HIFU treatment is expected to be less painful than other treatments used. The treatment is quick, and typically takes less than 1 minute for a each area the size of a typical neurofibroma.

ELIGIBILITY:
Inclusion Criteria:

* Males and females 18 years of age or older.
* Patients with a clinical diagnosis of NF1 based on germline genetic testing or by meeting the internationally recognized criteria given by the Clinical Care Advisory Board of the National Neurofibromatosis Foundation (now the Children's Tumor Foundation)
* Patients must be seeking active treatment for cNF.
* Patients must have ≥ 8 paired cNF that are visible and measure a minimum of 2 mm in size. These must be in areas amenable to treatment and surveillance.
* Patients with Fitzpatrick Type I to VI skin-type
* Able and willing to comply with all visits, treatments, evaluations, schedules, and requirements.
* Patients shall have received oral and written study information, accepted participation and signed the informed consent document.
* Patients who are willing and mentally and physically capable to understand and follow the treatment and follow-up schedule including post-treatment care instructions.
* Patients who are willing to have photographs and images taken of the treated lesions to be used anonymously or coded in evaluations and publications.

Exclusion Criteria:

* Patients who are undergoing other treatment modalities or investigational agents for their cNF lesions.
* Individuals who cannot give informed consent or adhere to study schedule.
* Patients who are actively tanning during the course of the study.
* Patients with adverse reactions to compounds of any external agent in use.
* Patients with known allergy to injectable anesthetics (relevant for biopsy only).
* Patients with any condition which, in the Investigator's opinion, would make it unsafe (for the participant or study personnel) to treat the participant as part of this research study.
* Patients, where target treatment may cause the acoustic beam to enter the eye.
* Pregnant females, due to possible discomfort with the procedure even though the procedure is localized and there is no new drug.
* Patients with tendency for keloid and hypertrophic scar formation .
* Patients with impaired wound healing.
* Patients with any other acute or chronic condition which, in the opinion of the investigator, could interfere with the conduct of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-04-13 (Actual); Primary Completion 2024-01-17 (Actual); Study Completion 2024-01-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- Bispebjerg Hospital, Copenhagen, Capital Region, Denmark
- Sahlgrenska University Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- TOOsonix System ONE-M: Cutaneous neurofibromas will be treated by high intensity focused ultrasound.
  TOOsonix System ONE-M: Selected neurofibromas will be treated by high intensity focused ultrasound.
  Untreated fibromas will be used for controls.
Period: Overall Study
Arm/Group | TOOsonix System ONE-M
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | TOOsonix System ONE-M
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Sweden | 10
  Denmark | 10

OUTCOME MEASURES:

1. Primary Outcome: Short Term Safety Profile - Adverse Events
Description: The grade of any adverse events (AE) requiring medical intervention within three months of treatment should be low. Device-based treatment will be considered tolerable if less than 30% of participants treated have an "Overall AE Score" larger than Grade 2 AE at the 3-month follow-up (visit 4).
  Measured by a grading scale based on Common Terminology Criteria for Adverse Events (CTCAE), U.S. Department of health and human services, Ver 5.0, Nov 27, 2017.
Time Frame: 3 months
Population: The grade of any adverse events (AE) requiring medical intervention within three months of treatment was measured.
Measure: Count of Participants; unit: Participants
Arm/Group | TOOsonix System ONE-M
Number analyzed (Participants) | 20
Participants
  Participants with an "Overall AE Score" larger than Grade 2 at the 3-month follow-up (visit 4). | 0
  Participants with an "Overall AE Score" of Grade 2 or below at the 3-month follow-up (visit 4). | 20

2. Primary Outcome: Long Term Safety Profile - Healing
Description: The rate and nature of spontaneous healing of the treated cNF lesion and any safety related event including potential wound formation and wound healing should be equivalent to expectations from alternative method(s). Safety evaluation includes rating of treatment-associated sequele by end of study, e.g. dyspigmentation and scarring and overall investigator rating compared to expectations.
  Measured on 5-point grading from Very Unsatisfied to Very Satisfied.
Time Frame: 9 months
Population: Tumor size was clinically assesed relative to baseline at the 9-month follow-up visit (visit 7). The assessment was based on tumor size alone, e.g. investigators assessment of width, elevation, and volume. <5: larger; 5: unchanged; 6-7: some reduction; 8-10: major reduction or no longer visible.
Measure: Number; unit: Tumors
Units Other Than Participants: Tumors
Arm/Group | TOOsonix System ONE-M
Number analyzed (Participants) | 20
Number analyzed (Tumors) | 92
Tumors
  Larger tumor size (<5) | 6
  Unchaged (5) | 16
  Some reduction (6-7) | 25
  Major reduction or no longer visible (8-10 | 45

3. Secondary Outcome: Long Term Safety Profile - Adverse Events
Description: Any objective adverse effect or event, local or systemic, related to the treatment and the investigational device.
  Measured by a grading scale based on Common Terminology Criteria for Adverse Events (CTCAE), U.S. Department of health and human services, Ver 5.0, Nov 27, 2017.
Time Frame: 9 months
Population: The grade of any adverse events (AE) requiring medical intervention within nine months of treatment was measured.
Measure: Count of Participants; unit: Participants
Arm/Group | TOOsonix System ONE-M
Number analyzed (Participants) | 20
Participants
  Participants with an "Overall AE Score" larger than Grade 2 at the 9-month follow-up (visit 7) | 0
  Participants with an "Overall AE Score" of Grade 2 or below at the 9-month follow-up (visit 7). | 20

ADVERSE EVENTS:
Time Frame: Participants recieved a single treatment with the investigational device. Follow-up was conducted after 1 week, 3 months, 6 months, and 9 months.
Description: The following criteria were used: U.S. Department of Health and Human Services. Common Terminology Criteria for Adverse Events (CTCAE). Version 5.0. Published online November 27, 2017. https://ctep.cancer.gov/protocoldevelopment/electronic_applications/docs/CTCAE_v5_Quick_Reference_5x7.pdf
Arm/Group | TOOsonix System ONE-M
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-15): https://cdn.clinicaltrials.gov/large-docs/82/NCT05119582/Prot_SAP_000.pdf